CLINICAL TRIAL: NCT00334425
Title: The Effect of LH-Priming During Early Follicular Phase on Ovarian Response and Pregnancy Outcome in GnRHa Down-Regulated Women, Stimulated With Exogenous Gonadotrophins in IVF Treatment
Brief Title: The Effect of LH-Priming During Early Follicular Phase in IVF Treatment.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Jutland Regional Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2005
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2006-06-13 (Estimated); Status verified 2006-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Menotropins; follitropin alfa

INTERVENTIONS:
Drug: MENOPUR; GONAL-F

SUMMARY:
To evaluate the effect of LH-activity supplementation during the early follicular phase in GnRHa down-regulated women undergoing IVF in terms of S-Estradiol levels on hCG day by comparing different combinations with HP-HMG and r-FSH.

ELIGIBILITY:
Inclusion Criteria:

* Females between the ages of 18- 38 years (both included) at the time of randomisation
* Patients for whom treatment with gonadotrophins and GnRH agonist (long protocol) in IVF setting is considered appropriate according to the criteria of the participating centre
* Infertility for at least 1 year before randomisation (except for tubal infertility)
* A maximum of two previous consecutive unsuccessful IVF cycles (i.e. not resulting in an ongoing pregnancy
* 25- 34 days of menstruation cycle
* Body mass index (BMI) < 29 kg/m2

Exclusion Criteria:

* Any clinically significant systemic disease (e.g., insulin dependent diabetes)
* Endocrine or metabolic abnormalities (pituitary, adrenal, thyroid, pancreas, liver, or kidney) which can compromise participation in the study
* Any concomitant medications that would interfere with evaluation of study medications. Specifically, any non-study hormonal therapy (except for thyroid medication), prostaglandin inhibitors (NSAIDs, including aspirin) and psychotropic agents (phenothiazine's, major tranquillisers) at the time of study entry. Note: these medications are disallowed for the study duration.
* Presence of clinically significant uterine fibroids
* Undiagnosed vaginal bleeding
* Tumours of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus
* Pregnancy, lactation or contraindication to pregnancy - must be confirmed by negative urinary pregnancy test at randomisation

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150
Dates: Start 2006-04

PRIMARY OUTCOMES:
Circulatory levels of Estradiol on the day of hCG

SECONDARY OUTCOMES:
Total number of follicles as well as the numbers of follicles <10mm, 10-14 mm, >14mm day during gonadotrophin treatment and at the end of stimulation prior to hCG injection
E2 per follicle >14 mm
Total number of oocytes retrieved
fertilization rate
serum hCG > 10 IU/l on day 12-14 after embryo transfer
implantation rate
transferable embryos
Clinical pregnancy rate
Ongoing pregnancy rate
embryo quality
Serum; LH, FSH, Androstenedione, Progesterone, hCG and Inhibin-B. Progesterone seven days after ET day
Intra follicular levels of; endocrine parameters
Endometrial thickness; hCG day (minus 0-2 days)
Total gonadotrophin dose administered

CONTACTS AND LOCATIONS:
Overall Officials: Peter Humaidan, M.D., Principal Investigator — Fertilitetsklinikken Sygehus Viborg
Locations (1):
- Fertilitetsklinikken Sygehus Viborg, Skive, Denmark